CLINICAL TRIAL: NCT05875571
Title: Intravenous Ketorolac Administration to Attenuate Post-procedural Pain Associated With Intrauterine Device Placement: A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Intravenous Ketorolac Administration to Attenuate Post-procedural Pain Associated With Intrauterine Device Placement
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Shahwar Yousuf, Principal Investigator, Pediatric Critical Care Fellow, Arkansas Children's Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 275563
Record Dates: First submitted 2023-05-08; First posted 2023-05-25 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: IUD; Healthy Female; Contraception; IUD Insertion Complication
MeSH Terms: interventions — Ketorolac; Ketorolac Tromethamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The provider and participant will be masked and will not know if the patient is getting the study drug or placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ketorolac (Active Comparator): The group of patients will receive IV Ketorolac before placement of IUD under sedation.
  Interventions: Drug: Ketorolac
- Placebo (Placebo Comparator): The group of patients will receive placebo before placement of IUD under sedation.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketorolac — Patients will get IV ketorolac during IUD placement under sedation
  Other Names: toradol
  Arms: Ketorolac
Drug: Placebo — Patients will get IV placebo during IUD placement under sedation
  Arms: Placebo

SUMMARY:
Intrauterine devices (IUDs) are a popular form of long-acting reversible contraception, with a high efficacy rate and few side effects. The insertion procedure for IUDs can be uncomfortable and painful. Sedation may be needed to improve patient comfort. The use of IUDs is increasing in the adolescent population, but perceived pain is a barrier to placement.

Propofol is a commonly used agent for pediatric procedural sedation, but it has no analgesic properties. Ketorolac, a nonsteroidal anti-inflammatory drug, has been shown to reduce pain in adults and improve patient satisfaction when used prior to IUD placement..

The current study aims to determine if ketorolac, given in combination with propofol for IUD placement in adolescents, can improve comfort during placement and reduce pain following the procedure. Enrolled patients will receive ketorolac or placebo, in addition to propofol, for IUD placement. By comparing the outcomes of these two groups of patients, we can gain a better understanding of the optimal approach to sedation for IUD insertion in adolescents.

DETAILED DESCRIPTION:
Background and Significance: IUDs are safe, effective, and reversible forms of contraception. They are available in two forms in the United States: non-hormonal (copper) and levonorgestrel hormonal devices. There are very few contraindications to placement and few associated side effects. Despite these facts, only 14% of women aged 15-44 currently use an IUD1. Data over recent years show an increase in IUD usage among younger women, and the American College of Obstetricians and Gynecologists (ACOG) support use in adolescent patients, many of which seek care from pediatric providers2. IUDs are easy to place and remove, with most procedures occurring in the office setting.

One barrier to more widespread use of IUDs may be the perception of pain associated with insertion, especially among younger patients. One study of 100 nulligravid women reported a 78% incidence of "moderate" or "severe" pain with IUD placement3. Several studies have evaluated various methods to attenuate the pain and anxiety associated with IUD placement, including behavioral interventions4, topical and injectable lidocaine applied to the cervix5,6, and injectable medications7. The ACOG currently recommends taking over-the-counter pain medications prior to IUD placement, though no specific medications are mentioned. Some adolescent patients require procedural sedation due to perceived pain, previous unsuccessful office procedures, developmental delay, and chronic pelvic pain, among other indications.

Ketorolac is a nonsteroidal anti-inflammatory drug (NSAID), available in oral and injectable forms. It is used for moderately severe pain, often after an operation or painful procedure. Time to onset of analgesia with injectable ketorolac (IV or IM) is approximately 30 minutes, with maximum effect at 1-2 hours, and a median duration of 6 hours. Ketorolac, given orally or as an intramuscular injection (IM), has been shown to effectively attenuate the pain associated with in-office placement of IUDs7,8. We hypothesize that the administration of IV ketorolac, given during sedation for IUD placement, will lead to a decrease in post-procedural pain.

Project Design and Methods: A randomized, double-blind, placebo-controlled trial will test the stated hypotheses associated with the specific aims above. All patients undergoing IUD placement under sedation, provided by the pediatric critical care sedation service at Arkansas Children's Hospital (ACH), will be eligible for enrollment. Patients meeting inclusion/exclusion criteria (see below) will be randomized to ketorolac or placebo after providing informed consent/assent. IUD placement will be performed by the pediatric gynecology service at ACH, using one of two levonorgestrel devices (Kyleena or Mirena). In addition to the study drug, propofol will be used for sedation. All subjects will be sedated with propofol in the following manner: 1mg/kg IV loading dose (10mg additional doses to achieve sedation), followed by a 150mcg/kg/min infusion rate during the procedure. Additional 10mg boluses will be given at the discretion of the seditionist (Pediatric Critical Care Medicine or Pediatric Emergency Medicine physician) and will be recorded for comparison as a secondary outcome measure.

Study Drug and Randomization Procedure: All eligible subjects will be randomized to ketorolac or placebo using simple randomization. A randomization schedule will be constructed using a random number generator. The study pharmacist will dispense ketorolac or placebo based on the randomization schedule. All study investigators and clinical staff will be blinded to group assignment. Ketorolac and placebo will be dispensed in identical syringes in identical volumes. Study drug will be administered intravenously by the sedation nurse at least 30 minutes prior to the start of sedation for IUD placement.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring sedated IUD placement at Arkansas Children's Hospital

Exclusion Criteria:

* Allergy to ketorolac or other NDSAID
* Known history of renal impairment
* History of GI bleeding of peptic ulcer disease

Ages: 13 Years to 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Female adolescent patients undergoing IUD placement
Enrollment: 18 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Comparison of Post procedural pain after IUD placement | 24 hours
  The primary outcome will be comparison of post-procedural pain using the Numerical Pain Rating Scale in ketorolac vs placebo group. The scale ranges from 0 to10 where 0 = no pain at all and 10= worst pain ever. Lower score indicates improvement in pain while a higher score indicates worsening of pain.

SECONDARY OUTCOMES:
number of propofol boluses required during sedation | 24 hours
total propofol dose (mg/kg) given in each group | 24 hours
  total propofol dose will be obtained from EHR and both groups will be compared for this purpose

CONTACTS AND LOCATIONS:
Locations (1):
- Arkansas Childrens Hospital, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jatlaoui TC, Riley HEM, Curtis KM. The safety of intrauterine devices among young women: a systematic review. Contraception. 2017 Jan;95(1):17-39. doi: 10.1016/j.contraception.2016.10.006. Epub 2016 Oct 19. PMID 27771475
- [Background] Hall AM, Kutler BA. Intrauterine contraception in nulliparous women: a prospective survey. J Fam Plann Reprod Health Care. 2016 Jan;42(1):36-42. doi: 10.1136/jfprhc-2014-101046. Epub 2015 Apr 8. PMID 25854550
- [Background] Lambert T, Truong T, Gray B. Pain perception with cervical tenaculum placement during intrauterine device insertion: a randomised controlled trial. BMJ Sex Reprod Health. 2020 Apr;46(2):126-131. doi: 10.1136/bmjsrh-2019-200376. Epub 2019 Oct 30. PMID 31666302
- [Background] Panichyawat N, Mongkornthong T, Wongwananuruk T, Sirimai K. 10% lidocaine spray for pain control during intrauterine device insertion: a randomised, double-blind, placebo-controlled trial. BMJ Sex Reprod Health. 2021 Jul;47(3):159-165. doi: 10.1136/bmjsrh-2020-200670. Epub 2020 Jun 26. PMID 32591417
- [Background] Mody SK, Farala JP, Jimenez B, Nishikawa M, Ngo LL. Paracervical Block for Intrauterine Device Placement Among Nulliparous Women: A Randomized Controlled Trial. Obstet Gynecol. 2018 Sep;132(3):575-582. doi: 10.1097/AOG.0000000000002790. PMID 30095776
- [Background] Ngo LL, Ward KK, Mody SK. Ketorolac for Pain Control With Intrauterine Device Placement: A Randomized Controlled Trial. Obstet Gynecol. 2015 Jul;126(1):29-36. doi: 10.1097/AOG.0000000000000912. PMID 26241253
- [Background] Crawford M, Davy S, Book N, Elliott JO, Arora A. Oral Ketorolac for Pain Relief During Intrauterine Device Insertion: A Double-Blinded Randomized Controlled Trial. J Obstet Gynaecol Can. 2017 Dec;39(12):1143-1149. doi: 10.1016/j.jogc.2017.05.014. Epub 2017 Aug 18. PMID 28826645
- [Background] Karcioglu O, Topacoglu H, Dikme O, Dikme O. A systematic review of the pain scales in adults: Which to use? Am J Emerg Med. 2018 Apr;36(4):707-714. doi: 10.1016/j.ajem.2018.01.008. Epub 2018 Jan 6. PMID 29321111
- [Background] Chaves IA, Baeta T, Dolabella GB, Barbosa LR, Almeida NM, Oliveira FR, Oliveira EC, L Silva-Filho A, Rocha ALL. Pain scores at the insertion of the 52 MG levonorgestrel-releasing intrauterine system among nulligravidas and parous women. Eur J Contracept Reprod Health Care. 2021 Oct;26(5):399-403. doi: 10.1080/13625187.2021.1925882. Epub 2021 Jun 7. PMID 34096433